CLINICAL TRIAL: NCT02289131
Title: Oral Care Intervention In Mechanically Ventilated Adults: Renewal
Brief Title: Frequency of Oral Care Intervention Study
Acronym: FOCIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Tampa General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO 00016479; 2R01NR007652-10A1 (NIH)
Record Dates: First submitted 2014-11-04; First posted 2014-11-13 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Respiratory Failure
Keywords: oral care
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Frequency of Once a Day (Experimental): Tooth Brushing Protocol to be provided at 8:00 am (+/- 1.5 hours)
  Interventions: Procedure: Tooth Brushing Protocol
- Frequency of Twice a Day (Experimental): Tooth Brushing Protocol to be provided at 8:00 am (+/- 1.5 hours) Tooth Brushing Protocol to be provided at 1:00 pm (+/- 1.5 hours)
  Interventions: Procedure: Tooth Brushing Protocol
- Frequency of Three Times a Day (Experimental): Tooth Brushing Protocol to be provided at 8:00 am (+/- 1.5 hours) Tooth Brushing Protocol to be provided at 1:00 pm (+/- 1.5 hours) Tooth Brushing Protocol to be provided at 6:00 pm (+/- 1.5 hours)
  Interventions: Procedure: Tooth Brushing Protocol

INTERVENTIONS:
Procedure: Tooth Brushing Protocol — A 2-minute tooth brushing protocol, followed by a mouthwash rinse and application of moisturizer for a total of approximately 15 minutes.

SUMMARY:
Tooth brushing for patients with breathing tubes is routinely provided by the bedside nurse as part of clinical care. The purpose of this study is to determine how often tooth brushing should occur for adult patients with breathing tubes (mechanical ventilation), balanced with equivalence and safety.

DETAILED DESCRIPTION:
A total of 345 adult subjects who are intubated and require mechanical ventilation will be randomly assigned to one of the three different tooth brushing frequency groups: once a day, twice a day or three times a day, up to a maximum of seven days. Teeth will be brushed with a soft child size toothbrush will take approximately 2 minutes. Following tooth brushing, the mouth will be rinsed with alcohol-free mouthwash and oral fluids will be removed with an oral suction tip. Moisturizing gel will be gently applied. The complete intervention requires approximately 15 minutes.

Information will be collected will include clinical condition, medications, age, gender, and smoking status. Once every day, digital pictures will be taken of each tooth (takes approximately five minutes) using a small intraoral camera to be evaluated for plaque by a dental hygienist that is blinded to frequency group assignment. Once every day, gingival crevicular fluid samples (takes 30 seconds) to look for factors that predict infection.

Gingival crevicular fluid samples and digital pictures of the teeth will also be collected on day 1, day 3 and day 5 after extubation.

ELIGIBILITY:
Inclusion Criteria:

* within 36 hours of initial intubation,
* have at least one tooth, and
* they or their legally authorized representative are able to provide informed consent in English or Spanish.

Exclusion Criteria:

* anticipation by the clinical provider of imminent patient death, or
* medical contraindication to tooth brushing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2014-12-31 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Dental Plaque as measured by University of Mississippi Oral Hygiene Index | Participants will be followed for the duration of the study, an expected average of 10 days.
  University of Mississippi Oral Hygiene Index
Gingival Inflammation as measured by Gingival Crevicular Fluid Samples | Participants will be followed for the duration of the study, an expected average of 10 days.
  Gingival Crevicular Fluid Samples

SECONDARY OUTCOMES:
Systemic Inflammatory Response Syndrome as measured by SIRS Criteria | Participants will be followed for the duration of the study, an expected average of 10 days.
  SIRS Criteria
Hospital Acquired Infection as measured by positive epidemiologic surveillance report for VAE (including VAP), bacteremia, sepsis | Participants will be followed for the duration of the study, an expected average of 10 days.
  positive epidemiologic surveillance report for Ventilator Associated Event (including VAP), bacteremia, sepsis
Length of Hospital Stay | Participants will be followed for the duration of hospital stay, an expected average of 10 days.
  Number of days from hospital admission date to hospital discharge date
Length of Intubation | Participants will be followed for the duration of the study, an expected average of 10 days.
  Number of days from intubation date to extubation date

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L Munro, PhD, Principal Investigator — University of Miami; Kevin E Kip, PhD, Principal Investigator — University of South Florida
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT02289131/Prot_SAP_000.pdf